CLINICAL TRIAL: NCT02980562
Title: Comparison of a Split Dose Bowel Preparation With 2-L Polyethylene Glycol Plus Ascorbic Acid and 1-L Polyethylene Glycol Plus Ascorbic Acid and Bisacodyl Prior to Colonoscopy
Brief Title: Comparison of Low Volume PEG-Asc and Lower Volume PEG-Asc With Bisacodyl
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Seung Hun Kang, Fellow, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Korea University preparation
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-11

CONDITIONS: Bowel Disease; Colon Adenoma
Keywords: Bowel preparation; Ascorbic acid; Bisacodyl; Polyethylene glycol
MeSH Terms: conditions — Intestinal Diseases | interventions — Polyethylene Glycols; Bisacodyl

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2L Polyethylene glycols-Asc (Active Comparator): 1 L of PEG containing ascorbic acid (PEG A) was taken at 8:00 pm on the day before the colonoscopy, followed by an extra 500 mL of water. The second 1-L of PEG containing ascorbic acid was taken 4 h before the colonoscopy examination, with an additional 500 mL of water. Each liter of preparation and the extra 500 mL water had to be consumed within 2 h of the procedure. All colonoscopies were performed between 9 am and 1 pm.
  Interventions: Drug: Polyethylene Glycols
- 1L PEG-Asc plus bisacodyl (Active Comparator): 10 mg bisacodyl at 9:00 pm on the day before the colonoscopy. Four hours before the colonoscopy examination, 1 L of PEG containing ascorbic acid was taken, followed by an additional 1 L of water. The preparation was completed 2 h before the examination. All colonoscopies were performed between 9 am and 1 pm.
  Interventions: Drug: Bisacodyl

INTERVENTIONS:
Drug: Polyethylene Glycols — (Split dose 2L PEG-Asc)
  Other Names: Coolprep®; Taejoon Pharmaceuticals, Seoul, Korea
  Arms: 2L Polyethylene glycols-Asc
Drug: Bisacodyl — (1L PEG-Asc plus bisacodyl)
  Other Names: Coolprep®; Taejoon Pharmaceuticals, Seoul, Korea; Dulcorax-S®; Boehringer Ingelheim, Seoul, Korea
  Arms: 1L PEG-Asc plus bisacodyl

SUMMARY:
Recently a low-volume polyethylene glycol containing ascorbic acid (PEG-Asc) formulation has proven as safe and effective as traditional 4-L PEG solutions for colonoscopy preparation. However, currently available aqueous purgative formulations are poorly tolerated. The aim of this study was to compare a split-dose 2-L PEG-Asc and a 1-L PEG-Asc with bisacodyl (10 mg) formulation to determine the quality of bowel cleansing and patient tolerability.

DETAILED DESCRIPTION:
- Study design A single center, randomized, comparative observer-blinded study was performed from May 2015 to September 2015 at the Department of Gastroenterology and Digestive Endoscopy at Korea University Anam Hospital (Seoul, Korea).

In total, 200 outpatients received lower volume 1-L PEG with ascorbic acid plus bisacodyl (1L-PEG/AB) or low volume 2-L PEG with ascorbic acid (2L-PEG/A) in a 1:1 ratio.

At the time of registration, subjects were randomly allocated to either group. They were randomized by a computer-generated list and were provided with written instructions. All patients provided written informed consent.

* Patients All patients between the ages of 20 and 75 years. Patients were excluded from the analysis if they had known or suspected gastrointestinal obstruction, Ileus, severe heart failure, uncontrolled hypertension (systolic pressure > 170 mmHg, diastolic pressure > 100 mmHg), severe constipation, clinically significant electrolyte abnormalities, any prior bowel resection, or significant gastroparesis.
* Bowel preparation In the 2L-PEG/A group, 1 L of PEG containing ascorbic acid was taken at 8:00 pm on the day before the colonoscopy, followed by an extra 500 mL of water. The second 1-L of PEG containing ascorbic acid was taken 4 h before the colonoscopy examination, with an additional 500 mL of water. Each liter of preparation and the extra 500 mL water had to be consumed within 2 h of the procedure.

The 1L-PEG/AB group received 10 mg bisacodyl at 9:00 pm on the day before the colonoscopy. Four hours before the colonoscopy examination, 1 L of PEG containing ascorbic acid was taken, followed by an additional 1 L of water. The preparation was completed 2 h before the examination. All colonoscopies were performed between 9 am and 1 pm.

- Assessment by endoscopists Colonoscopies were performed by two expert endoscopists who were blinded to the preparation regimen. These two endoscopists worked for more than 5 years at our institution.

Bowel cleansing was scored by the same endoscopist performing the colonoscopy. To assess the cleansing quality of the bowel preparations, the Boston Bowel Preparation Scale (BBPS) and the Aronchick Bowel Preparation Scale (ABPS) were used.

- Assessment of patient tolerability and adverse events Before the colonoscopy procedure, patients completed questionnaires about their symptoms associated with the preparations to assess tolerability. Patients were asked to assess the degree of abdominal fullness, abdominal pain, nausea, vomiting, sleep disturbances, and general discomfort using a 5-point scale (i.e., none, mild, moderate, severe, or very severe).

The palatability of the preparation was graded in 5 categories: very good, good, acceptable, disgusting, and bad.

- Sample size and statistical analysis A sample size of at least 89 patients group was required for each treatment group to detect a difference in treatment success of a 5% type-I error rate and 80% power for a two-tailed χ2 test. Our sample size was based on the results from a pilot study that was conducted in our hospital and included 35 patients in each group. It was estimated that the efficacy for excellent treatment success would be 49% with PEG-2L/A and 30% with PEG-1L/AB. Based on these data, we decided to collect 100 patients per treatment group for study.

Continuous variables were expressed as mean ± standard deviation (SD), and discontinuous variables were expressed as counts and percentages. SPSS 20.0 for Windows (SPSS Inc., Chicago, IL, US) was used for data entry and statistical analyses. For the analyses between the two treatment groups, Students t-test as appropriate was used to compare continuous variables and either the Chi-square or Fisher's exact test were used for categorical data. The p-values < 0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* All patients between the ages of 20 and 75 years who were scheduled to undergo colonoscopy

Exclusion Criteria:

* aged more than 75 years.
* known or suspected gastrointestinal obstruction, Ileus
* severe heart failure
* uncontrolled hypertension (systolic pressure > 170 mmHg, diastolic pressure > 100 mmHg)
* severe constipation
* clinically significant electrolyte abnormalities
* any prior bowel resection, or significant gastroparesis.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The quality of the bowel preparation using preparation scale | 20 minutes
  Preparation scale

SECONDARY OUTCOMES:
The patient's tolerability | 30 minutes before the colonoscopy
  Patients were asked with questionnaires about the symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Yoon Tae Jeen, Study Director — Division of Gastroenterology and Hepatology, Department of Internal Medicine, Institute of Gastrointestinal Medical Instrument Research, Korea University College of Medicine; Seung Hun Kang, Principal Investigator — Division of Gastroenterology and Hepatology, Department of Internal Medicine, Institute of Gastrointestinal Medical Instrument Research, Korea University College of Medicine

REFERENCES:
- [Derived] Kang SH, Jeen YT, Lee JH, Yoo IK, Lee JM, Kim SH, Choi HS, Kim ES, Keum B, Lee HS, Chun HJ, Kim CD. Comparison of a split-dose bowel preparation with 2 liters of polyethylene glycol plus ascorbic acid and 1 liter of polyethylene glycol plus ascorbic acid and bisacodyl before colonoscopy. Gastrointest Endosc. 2017 Aug;86(2):343-348. doi: 10.1016/j.gie.2016.10.040. Epub 2016 Nov 23. PMID 27889546